CLINICAL TRIAL: NCT05009459
Title: eVISualisation of Physical Activity and Pain (eVIS) for Patients With Chronic Pain Participating in Swedish Interdisciplinary Pain Rehabilitation Programs: a Registry-based Randomized Controlled Clinical Trial
Brief Title: eVISualisation of Physical Activity and Pain (eVIS) for Patients With Chronic Pain
Acronym: eVIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Linda Vixner, Docent in Medical Sciences/Deputy Head of Research Centre for Public Health and Sports (RePS), Dalarna University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00491
Record Dates: First submitted 2021-06-29; First posted 2021-08-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain
Keywords: Chronic pain Registry-based randomized clinical trial
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eVIS + Treatment as usual (interdisciplinary pain rehabilitation program) (Experimental): Participant takes part of the unit´s program with an addition of eVIS. eVIS consists of objectively measured physical activity tracking using a wrist-worn activity tracker (Fitbit Versa 2) is combined with a daily activity goal (steps/day) and daily patient reports of known important clinical outcome assessments: pain intensity and its affect on daily activities and pharmaceutical consumption. Data is collected and visualized in a purpose-developed web application, Pin And TRaining ON-line (PATRON), which can be used by the patient and the IPRP-team to follow and adjust individual physical activity levels.
  Interventions: Behavioral: eVIS
- Treatment as usual (interdisciplinary pain rehabilitation program) (No Intervention): Participant takes part of the unit´s program with an addition of daily self-report of pain intensity (0-10), affect of pain on daily activities (0-10), and pharmacological consumption.

INTERVENTIONS:
Behavioral: eVIS — To facilitate individualized physical activity levels within the Swedish IPRP setting, an eVISualisation (eVIS) of physical activity and pain intervention has been systematically developed. eVIS is designed to target facilitating mechanisms for behavior change, such as outcome expectations, self-monitoring, self-evaluation, and self-efficacy, which are theoretically framed by the Social Cognitive Theory by Bandura. In eVIS, objectively measured physical activity tracking using a wrist-worn activity tracker (Fitbit Versa 2) is combined with a daily activity goal (steps/day) and daily patient reports of known important clinical outcome assessments: pain intensity and its affect on daily activities30-34 and pharmaceutical consumption. Data is collected and visualized in a purpose-developed web application, Pin And TRaining ON-line (PATRON), which can be used by the patient and the IPRP-team to follow and adjust individual physical activity levels.
  Arms: eVIS + Treatment as usual (interdisciplinary pain rehabilitation program)

SUMMARY:
Introduction: Living with chronic pain often involves negative consequences. Interdisciplinary Pain Rehabilitation Programs (IPRPs), a subset of Interdisciplinary Treatment (IDT) includes physical activity and exercise and is considered superior to single-treatment measures in patients with chronic pain. However, effects emerge sub-optimal and as many as 30% of patients deteriorate in some outcomes. A novel intervention, eVISualisation (eVIS) of physical activity and pain, has been systematically developed to facilitate patients in reaching and maintaining recommended individualized physical activity levels. The aim is to transparently report on methodology, outcome assessments, and processes for a registry-based randomized controlled trial (R-RCT) initiated as an internal pilot study.

Methods and analysis: The R-RCT will recruit approximately 400 patients with chronic pain who are registered at primary and specialized IPRP units (n=15) in Sweden. Participants will be randomly allocated to either an IPRP + eVIS or the control group that will receive only IPRP treatment. eVIS entails objectively measured physical activity (steps) and patient-reported outcomes (pain intensity, affect on daily activities, pharmaceutical consumption) collected and visualized in the web application PATRON. Data from an initial 30 participants completing the study period (6 months) will be included in a pilot study designed to evaluate recruitment- and randomization processes, standardized effect size, sample size, characteristics of outcomes, follow-up rates of the R-RCT. Outcome variables will be extracted from PATRON and from six national registries. Multivariate statistics and repeated measures analyses will be performed. Quality Adjusted Life Years (QALYs) and Incremental Cost Effectiveness Ratio (ICER) will be calculated for cost effectiveness evaluation.

Ethics/dissemination: The Swedish Ethics Review Board granted approval (Dnr 2021/02109). Results will be disseminated through peer-review journals.

ELIGIBILITY:
Inclusion Criteria:

Swedish IPRP treatment criterias will be applied as patients entering the trial must be accepted for IPRP: Principal IPRP inclusion criteria are:

* persistent or intermittent pain lasting ≥3 months
* pain affecting daily activities to a large extent,
* completed systematic assessment and non-pharmacological optimization is completed,
* screening for psychosocial risk factors and differential diagnosis completed

In addition the following criterias will be appled:

* Patients aged 18-67 years.
* Patients must be able to hear, see, and comprehend spoken and written Swedish
* Daily access to a computer, smartphone, or tablet.

Exclusion Criteria:

* Patients who need to use a walking aid indoors.
* Patients living with pain caused by systemic disease or malignancies.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical health | 12 months follow up after IPRP
  Physical health domain by RAND-36, ranging from 0 to 100, with high values indicating good health.

SECONDARY OUTCOMES:
Physical and mental health | 6, 24, 36 months after IPRP
  RAND-36 health survey, ranging from 0 to 100, with high values indicating good health.
Objectively measured physical activity levels | Data will be collected daily during study period (6 months)
  Steps per day collected by Fitbit Versa 2 synchronized to web application PATRON
Pain intensity last 24 hours | Data will be collected daily during study period (6 months)
  Pain intensity ("rate your average pain during the last 24 hours") by the Numeric Rating Scale (NRS), ranging from 0-10 with high values indicating high levels of pain. The scale is incorporated in the web application PATRON.
Pain interference | Data will be collected daily during study period (6 months)
  Data on self percieved pain interference on daily activities will be collected daily during study period ("rate how much your daily activities are affected by pain"). The scale is ranging from 0-10 with high values indicating high levels of interference. The scale is incorporated in the web application PATRON.
Drug name | Data will be collected daily during study period (6 months)
  Daily self reported data on drug name in the web application PATRON.
Drug dose | Data will be collected daily during study period (6 months)
  Daily self reported data on drug dose (example: 2 tablets per day) in the web application PATRON.
Drug strenght | Data will be collected daily during study period (6 months)
  Daily self reported data on drug strenght (example: 500 mg/tablet) in the web application PATRON.
Drug form | Data will be collected daily during study period (6 months)
  Daily self reported data on drug form (example: tablet, injection) in the web application PATRON.
Work form | 12 months follow up after IPRP
  Data on work form will be collected from Swedish national quality registry for pain rehabilitation.
Work extension | 12 months follow up after IPRP
  Data on work extension will be collected from Swedish national quality registry for pain rehabilitation.
Education level | 12 months follow up after IPRP
  Demografic data on the dispursion of education level (elementary, gymnasium, university, other) will be collected from Swedish national quality registry for pain rehabilitation
Pain intensity last seven days | 12 months follow up after IPRP
  Pain intensity ("rate your average pain during the last 7 days") will be measured daily using the Numeric Rating Scale (NRS) ranging from 0-10, with high values indicating high levels of pain. Collected through SQRP-PC and SQRP-SC
Pain regions | 12 months follow up after IPRP
  Patients' ratings on a form with 36 anatomical predefined areas (18 on the left side, 18 on the right side: 1) head/face, 2) neck, 3) shoulder, 4) upper arm, 5) elbow, 6) forearm, 7) hand, 8) anterior aspect of chest, 9) lateral aspect of chest, 10) belly, 11) genitals, 12) upper back, 13) lower back, 14) hip/gluteal area, 15) thigh, 16) knee, 17) lower leg, and 18) foot collected through SQRP-PC and SQRP-SC.
  Higher number of regions represents higher number of painful body regions .
Pain duration | 12 months follow up after IPRP
  Days. Collected through SQRP-PC and SQRP-SC. High number of days represents longer pain duration.
Self-rated mental health | baseline, 6, 12, 24 months follow up after IPRP.
  Data will be collected by the RAND-36 health survey collected through SQRP-SC and through email administered surveys. Values are ranging from 0 to 100, with high values indicating good mental health.
Self-rated health | baseline, 12, 24 months follow up after IPRP.
  Data will be collected by the EuroQol-5 dimensions (EQ-5D)The Swedish version of the EuroQol-5 dimensions, (3 level version) collected routinely in SQRP-PC and SQRP-SC. The first part of EQ-5D-3L consists of a descriptive system of 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with 3 severity levels (no/some/extreme problems). The 5 dimensions can be converted into a summary index (EQ-5D Index), which ranges from
  -0.594 to 1, where 1 represents "perfect health" and values below zero represent states "worse than death".
Physical activity | 12 months follow up after IPRP
  Data will be collected through SQRP-PC using the National Board of Health and Welfare's question on physical activity (0 - >300 minutes/week),The outcome represents minutes spent in physical activity/week. High values represents high level of physical activity,
Exercise | 12 months follow up after IPRP
  Data will be collected through SQRP-PC using the National Board of Health and Welfare's question on exercise (0 - >120 minutes/week)The outcome represents minutes spent in exercise. High values represents high level of exercise/week. .
Sedentary activities | 12 months follow up after IPRP
  Data will be collected through SQRP-PC using the National Board of Health and Welfare's question on, and sedentary behavior (0 - 15 hours/day).The outcome represents minutes spent in sedentary activities/week. High values represents high level of sedentary behavior.
Strenous exercise | 12 months follow up after IPRP
  In SQRP-SC, data is collected by the Godin-Shepard leisure-time physical activity questionnaire (number of times/week that strenuous exercise is performed). High values represents high levels of strenuous exersise per week.
Moderate exercise | 12 months follow up after IPRP
  In SQRP-SC, data is collected by the Godin-Shepard leisure-time physical activity questionnaire (number of times/week that moderate exercise is performed). High values represents high levels of moderate exersise per week.
Light exercise | 12 months follow up after IPRP
  In SQRP-SC, data is collected by the Godin-Shepard leisure-time physical activity questionnaire (number of times/week that light exercise is performed). High values represents high levels of light exersise per week.
Overall emotional distress | 12 months follow up after IPRP
  Data will be collected by the Hospital Anxiety and Depression Scale (HADS) in both SQRP-PC and SQRP-SC. HADS is a 14-item self-assessment questionnaire in which 7 items address anxiety and 7 items address depression (subscales; HADS-D - depression and HADS-A - anxiety).
  The subscale scores can range from 0 to 21, with lower scores indicating better function.
Pain catastrophizing | 12 months follow up after IPRP
  Data will be collected by the Pain Catastrophizing Scale (PCS) in both SQRP-PC and SQRP-SC. The PCS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52. Higher values indicating higher levels of catastrophizing
Psychosocial consequences - Pain intensity | 12 months follow up after IPRP
  Data will be collected by the Multidimensional Pain Inventory Scale Swedish version (MPI-S) in both SQRP-PC and SQRP-SC. The construct "psychosocial consequences" is measured by five subscales (total 22 items) where "pain intensity" is the first. The subscales and the index range from 0-6, with higher scores indicating better function.
Psychosocial consequences - Interference | 12 months follow up after IPRP
  Data will be collected by the Multidimensional Pain Inventory Scale Swedish version (MPI-S) in both SQRP-PC and SQRP-SC. The construct "psychosocial consequences" is measured by five subscales (total 22 items) where "interference" is the the second subscale. The subscales and the index range from 0-6. In "interference" higher scores indicate higher interference.
Psychosocial consequences - Life control | 12 months follow up after IPRP
  Data will be collected by the Multidimensional Pain Inventory Scale Swedish version (MPI-S) in both SQRP-PC and SQRP-SC. The construct "psychosocial consequences" is measured by five subscales (total 22 items) where "life control" is the third subscale. The subscales and the index range from 0-6, with higher scores indicating better function.
Psychosocial consequences - Affective distress | 12 months follow up after IPRP
  Data will be collected by the Multidimensional Pain Inventory Scale Swedish version (MPI-S) in both SQRP-PC and SQRP-SC. The construct "psychosocial consequences" is measured by five subscales (total 22 items) where "affective distress" is the fourth subscale. The subscales and the index range from 0-6, with higher scores indicating better function.
Psychosocial consequences - Social support | 12 months follow up after IPRP
  Data will be collected by the Multidimensional Pain Inventory Scale Swedish version (MPI-S) in both SQRP-PC and SQRP-SC. The construct "psychosocial consequences" is measured by five subscales (total 22 items) where "social support" is the fitth subscale. The subscales and the index range from 0-6, with higher scores indicating better function.
Pain acceptance | 12 months follow up after IPRP
  Will be collected in SQRP-PC using the Chronic Pain and Acceptance Questionnaire (CPAQ-8). The items on the CPAQ are rated on a 7-point scale from 0 (never true) to 6 (always true). Higher scores indicate higher levels of acceptance.
Life satisfaction | 12 months follow up after IPRP
  Will be collected by the Life Satisfaction Scale (LiSat) in both SQRP-PC and SQRP-SC. Each item is scored on a 6-point scale from 1 (very dissatisfied) to 6 (very satisfied). High values represents higher perceived life satisfaction.
Work ability | 12 months follow up after IPRP
  Will be collected by the Work Ability Index (WAI) in SQRP-SC only. The scale ranges from 0 ("cannot work at all) to 10 (my ability to work is at its best right now) where higher levels indicate higher levels of work ability
Functional levels | 12 months follow up after IPRP
  Data on functional level will be collected by the Functional Rating Scale (FRI) ranging from 0-4 in each item, total score is 40 and high values represents highly affected functional levels. FRI is collected in SQRP-SC only
Sleep quality | 12 months follow up after IPRP
  Data on sleep quality will be collected by the Insomnia Severity Index (ISI) in SQRP-SC.
  The index consists of 10 items with response scale 0 (no difficulities) to 4 (major difficulities). High values represents major sleep difficulties.
Reasons for Sick leave | 12 months follow up after IPRP
  Demographic data on reasons for sick leave will be retrieved from the Swedish Social Insurance Agency's registry.
Sickness benefit | 12 months follow up after IPRP
  Data on sickness benefit (days and hours) during the study period will be retrieved from the Swedish Social Insurance Agency's registry
Days in work before new sick leave period | 12 months follow up after IPRP
  Data on days in work (partial or full time) per month in total before new sick leave period will be retrieved from the Swedish Social Insurance Agency's registry
Total sick leave | 12 months follow up after IPRP
  Data on length of total sick leave during the study period will be retrieved from the Swedish Social Insurance Agency's registry
Diagnosis | 12 months follow up after IPRP
  Demographic data on the incidence of diagnoses will be retrieved from the Patient registry.
Total number of days in care | 12 months follow up after IPRP
  Data on total number of days in care) will be retrieved from the Patient registry.
Quality Adjusted Life Years | 12 months follow up after IPRP
  The outcome will be calculated as Quality Adjusted Life Years (QALYs) which is a "utility value" that ranges between 1 (perfect health), and 0 = death. The standard treatment will be used as baseline and the calculation is a cost effectiveness calculation. Data on health-related quality of life will be used. Higher values of QALYs represents higher cost effectiveness of the intervention.
  The calculation formula is as follows: Years of Life x Utility Value = #QALYs
Defined pharmaceutical doses per day | 12 months follow up after IPRP
  Retrieved data from the Pharmaceutical registry will provide information on prescribed and collected pharmaceutical defined doses per day (DDD) which includes names, doses, sizes that have been collected from pharmacies, their costs, and whether the pharmaceutical is included in the subsidized pharmaceutical program.
Pharmaceutical costs | 12 months follow up after IPRP
  Retrieved data from the Pharmaceutical registry will provide information on costs of prescribed and collected pharmaceuticals in SEK.
Income | 12 months follow up after IPRP
  Data on disposable and earned income (SEK) as well as net income will be retrieved from the Income and taxation registry. High values represents high income.
Education | 12 months follow up after IPRP
  From the Population registry, data on education level and education orientation (focus) in addition to limited demographic data (sex, age) will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Vixner, Dr, Principal Investigator — School Health and Welfare
Locations (1):
- Dalarna University, Falun, Sweden

IPD SHARING:
Plan to Share IPD: Yes
.For all data generated during this project, the standards and guidelines set by the International Committee of Medical Journal Editors, will be followed. In detail, this statement implies the following:
  1. Results from research conducted under this project will be shared and disseminated by submission for publication in high-quality peer-reviewed journals, following relevant public access guidelines. In addition, findings will be presented at relevant international and national conferences.
  2. Deidentified individual data used in publications will be made available on reasonable request to principal investigator after completion of the trial, at the earliest 2024-01-01. However, such request must lie within the limits of the ethical approval for this project. In addition, to uphold data safety and other legal aspects relevant agreements must be established prior to data being available outside the research group.
  3. Supporting files will be available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For deidentifed individual data used in publications: start date 2024-01-01. For additional files (supporting information): start date 2022-03-01.
Access Criteria: Any data request must lie within the limits of the ethical approval for this project. In addition, to uphold data safety and other legal aspects relevant agreements must be established prior to data being available outside the research group.

REFERENCES:
- [Background] Sjoberg V, Westergren J, Monnier A, Lo Martire R, Hagstromer M, Ang BO, Vixner L. Wrist-Worn Activity Trackers in Laboratory and Free-Living Settings for Patients With Chronic Pain: Criterion Validity Study. JMIR Mhealth Uhealth. 2021 Jan 12;9(1):e24806. doi: 10.2196/24806. PMID 33433391
- [Background] Sjoberg V, Tseli E, Monnier A, Westergren J, LoMartire R, Ang BO, Hagstromer M, Bjork M, Vixner L. Effectiveness of the eVISualisation of physical activity and pain intervention (eVIS) in Swedish Interdisciplinary Pain Rehabilitation Programmes: study protocol for a registry-based randomised controlled clinical trial. BMJ Open. 2022 Apr 15;12(4):e055071. doi: 10.1136/bmjopen-2021-055071. PMID 35428627
- [Background] Tseli E, Sjoberg V, Bjork M, Ang BO, Vixner L. Evaluation of content validity and feasibility of the eVISualisation of physical activity and pain (eVIS) intervention for patients with chronic pain participating in interdisciplinary pain rehabilitation programs. PLoS One. 2023 Mar 10;18(3):e0282780. doi: 10.1371/journal.pone.0282780. eCollection 2023. PMID 36897847